CLINICAL TRIAL: NCT00905996
Title: A Randomized Controlled Trial Comparing Cyanoacrylate Injection Versus Beta-Blockers Versus No Treatment for Primary Prophylaxis of Gastric Variceal Bleed
Brief Title: Primary Prophylaxis of Gastric Varix Bleed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr S K Sarin, Department of Gastroenterology, G B Pant Hospital, New Delhi, India
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: SRM04
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Adhesives; Adrenergic beta-Antagonists; Propranolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endoscopic Cyanoacrylate injection (Active Comparator): Endoscopic injection of cyanoacrylate in the gastric varix until obturation
  Interventions: Procedure: Endoscopic cyanoacrylate injection
- No Intervention (No Intervention): No treatment offered for gastric varix
- Beta-blocker (propranolol) (Other): Beta-blocker (propranolol) was started at a dose of 20 mg twice daily. The principle of incremental dosing was used to achieve the target heart rate for propranolol. The dose was increased every alternate day to achieve a target heart rate of 55/min or to the maximal dose to 360 mg/day if the medication was well tolerated and the systolic blood pressure was > 90 mm Hg. On the occurrence of intolerable adverse effects, systolic blood pressure < 90 mm Hg or pulse rate < 55/min, the dose of the medication was decreased step-wise, and eventually stopped if these adverse events persisted. Reintroduction of the medication was attempted if cessation of the medication did not result in improvement of the reported side-effect.
  Interventions: Drug: Beta-blocker (propranolol)

INTERVENTIONS:
Procedure: Endoscopic cyanoacrylate injection — Endoscopic cyanoacrylate injection in gastric varix
  Other Names: Glue injection in gastric varix
  Arms: Endoscopic Cyanoacrylate injection
Drug: Beta-blocker (propranolol)
  Arms: Beta-blocker (propranolol)

SUMMARY:
In patients who have never bled from gastric varix (GOV2 and IGV1), cyanoacrylate injection will be better than both beta-blocker therapy and no treatment in prevention of gastric variceal bleed. The investigators conducted a randomized controlled trial in patients with gastric varix (GOV2 and IGV1) who never bled before, to study the efficacy of treatment with cyanoacrylate injection versus beta-blocker versus no treatment in prevention of first bleed from gastric varices.

DETAILED DESCRIPTION:
Patients are followed up every 3 months or at the time of end point or complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GOV2 with eradicated esophageal varix or IGV1, who had never bled from gastric varix were included.

Exclusion Criteria:

* Only esophageal varix, GOV1 with GOV2, acute bleed or past history of bleed from gastric varix, contraindications to beta-blocker therapy and cyanoacrylate injection.
* Prior injection of cyanoacrylate or sclerotherapy or variceal ligation or transjugular intrahepatic portosystemic shunt or balloon-occluded retrograde transvenous obliteration or balloon-occluded endoscopic injection sclerotherapy of gastric varix for prevention of bleeding from GV
* Patients already on beta-blocker or nitrates
* Undetermined origin of bleeding from esophageal varix or gastric varix
* Hepatic encephalopathy grade III/IV
* Hepatorenal syndrome
* Hepatocellular carcinoma
* Presence of deep jaundice (serum bilirubin > 10 mg/dl)
* Uremia
* Cerebrovascular accident
* Cardiorespiratory failure
* Pregnancy and patients not giving informed consent for endoscopic procedures

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Bleeding from gastric varix or death | Within 2 years

SECONDARY OUTCOMES:
Increase or decrease in the size of gastric varices, appearance of new esophageal varices and appearance or worsening of portal hypertensive gastropathy (PGP), complications | Within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — G B Pant Hospital, New Delhi, India
Locations (1):
- Shiv K Sarin, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Mishra SR, Sharma BC, Kumar A, Sarin SK. Primary prophylaxis of gastric variceal bleeding comparing cyanoacrylate injection and beta-blockers: a randomized controlled trial. J Hepatol. 2011 Jun;54(6):1161-7. doi: 10.1016/j.jhep.2010.09.031. Epub 2010 Nov 5. PMID 21145834